CLINICAL TRIAL: NCT03201263
Title: PRessure suppOrT vEntilation + Sigh in aCuTe hypoxemIc respiratOry Failure patieNts (PROTECTION): a Pilot Randomized Controlled Trial
Brief Title: Sigh in Acute Hypoxemic Respiratory Failure
Acronym: PROTECTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: European Society of Intensive Care Medicine (Other); University of Milan (Other); University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sigh study
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome; Ventilator Lung
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome | interventions — SigH protein, bacteria; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial, 2 groups, 1:1 randomisation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSV group (Active Comparator): Will be treated by standard of care for patients undergoing assisted mechanical ventilation (e.g., protective PSV settings, protocolized weaning, etc.).
  Interventions: Procedure: Standard of care
- PSV+Sigh group (Experimental): Will be treated by standard of care for patients undergoing assisted mechanical ventilation (e.g., protective PSV settings, protocolized weaning, etc.) + Sigh (short cyclic recruitment breath once every minute) until death or spontaneous breathing trial and extubation.
  Interventions: Procedure: Sigh

INTERVENTIONS:
Procedure: Sigh — Application of cyclic pressure control breath delivered at 30 cmH2O for 3 seconds once per minute in patients undergoing pressure support ventilation
  Other Names: Short cyclic recruitment breath
  Arms: PSV+Sigh group
Procedure: Standard of care — Standard of care
  Arms: PSV group

SUMMARY:
Mortality of intubated acute hypoxemic respiratory failure (AHRF) and acute respiratory distress syndrome (ARDS) patients remains considerably high (around 40%) (Bellani 2016). Early implementation of a specific mechanical ventilation mode that enhances lung protection in patients with mild to moderate AHRF and ARDS on spontaneous breathing may have a tremendous impact on clinical practice.

Previous studies showed that the addition of cyclic short recruitment maneuvers (Sigh) to assisted mechanical ventilation: improves oxygenation without increasing ventilation pressures and FiO2; decreases the tidal volumes by decreasing the patient's inspiratory drive; increases the EELV by regional alveolar recruitment; decreases regional heterogeneity of lung parenchyma; decreases patients' inspiratory efforts limiting transpulmonary pressure; improves regional compliances. Thus, physiologic studies generated the hypothesis that addition of Sigh to pressure support ventilation (PSV, the most common assisted mechanical ventilation mode) might decrease ventilation pressures and FiO2, and limit regional lung strain and stress through various synergic mechanisms potentially yielding decreased risk of VILI, faster weaning and improved clinical outcomes.

The investigators conceived a pilot RCT to verify clinical feasibility of the addition of Sigh to PSV in comparison to standard PSV.

The investigators will enrol 258 intubated spontaneously breathing patients with mild to moderate AHRF and ARDS admitted to the ICU.

Patients will be randomized through an online automatic centralized and computerized system to the following study groups (1:1 ratio):

* PSV group: will be treated by protective PSV settings until day 28 or death or performance of spontaneous breathing trial (SBT);
* PSV+Sigh group: will be treated by protective PSV settings with the addition of Sigh until day 28 or death or performance of spontaneous breathing trial (SBT).

Indications on ventilation settings, weaning, spontaneous breathing trial and rescue treatment will be specified.

DETAILED DESCRIPTION:
Steering committee: Tommaso Mauri, Laurent Brochard, Jean-Michel Constantin, Giuseppe Foti, Claude Guerin, Jordi Mancebo, Paolo Pelosi, Marco Ranieri, Antonio Pesenti Statistical support: Carla Fornari and Sara Conti

Specific aims

This pilot RCT will serve to test the hypothesis that application of PSV+Sigh in spontaneously breathing intubated patients with mild to moderate AHRF and ARDS is feasible and to collect preliminary data on the safety of such an approach.

Methods

Study design. The investigators will conduct a pilot RCT on intubated spontaneously breathing patients with mild to moderate AHRF and ARDS admitted to the ICU.

Ethics approval. The investigators will seek approval from the institutional review boards of each participating center prior to start of enrollment and consent/information will be obtained from each patient or next of kin following local regulations.

Prevalence of Sigh responders. After enrollment, FiO2 will be titrated to obtain SpO2 of 90-96% and then each patient will first undergo a clinical test of PSV vs. PSV+Sigh to assess the prevalence of Sigh responders vs. non-responders in respect to improved oxygenation. After 30 minutes of clinical PSV+Sigh, SpO2/FiO2 ratio will be collected again to quantify the number of patients in whom it increased (i.e., "Sigh responders").

Randomization. After this test, patients will be randomized through an online automatic centralized and computerized system to the following study groups (1:1 ratio):

* PSV group: will be treated by protective PSV settings until day 28 or death or performance of spontaneous breathing trial (SBT);
* PSV+Sigh group: will be treated by protective PSV settings with the addition of Sigh until day 28 or death or performance of spontaneous breathing trial (SBT).

PSV group settings. Initially, clinicians will set PSV to meet the following targets: tidal volume (Vt) of 6-8 mL/Kg of predicted body weight (PBW), with respiratory rate (RR) 20-35 bpm. In presence of Vt >8 ml/kg PBW and/or RR <20 bpm, PSV zero (CPAP) will be selected. FiO2 will be left as selected before the pre-randomization Sigh test, while PEEP will be left as clinically set.

PSV+Sigh group settings. Similarly, PSV in this group will be set with the same protective targets of the PSV group (see above) and cyclic pressure control phase at 30 cmH2O for 3 seconds delivered once per minute (i.e., Sigh) will be added. PSV+Sigh is an easy to implement ventilation mode and, for the present study, the investigators will use high performance ICU ventilators already available in each clinical unit. Briefly, ventilators will be switched to biphasic positive airway pressure mode (e.g., BiPAP on Drager ventilators, SIMV-PC on Maquet and GE, DuoPAP on Hamilton) with the lower pressure level set at clinical PEEP and the higher pressure level set at 30 cmH2O with a 3-second inspiratory time and then a 57-second expiratory time. This Sigh rate of one per minute can be obtained by virtually all the already available high performance ICU ventilators, thus, even though a lower Sigh rate might be regarded as more physiological, we choose the 1/min rate for feasibility and costs related to the future large RCT. FiO2 will be left as selected before the pre-randomization Sigh test.

Adjusting ventilation settings. In both groups, PSV will be adjusted at least every 8 hours in the following way:

* PSV support will be decreased by 2 cmH2O step if Vt >8 ml/kg PBW and/or RR <20;
* PSV support will be increased by 2 cmH2O step if Vt <6 ml/kg PBW and/or RR >35 and or signs of respiratory distress (e.g., marked use of the accessory muscles).
* PEEP and then FiO2 will be increased by 2 cmH2O and 0.1 steps if SpO2 is <90%;
* FiO2 and then PEEP will be decreased by 0.1 and 2 cmH2O steps if SpO2 is >96%; Sigh settings instead will be left unchanged until day 28, death or SBT.

Switch to controlled mechanical ventilation. In both groups, switch to protective controlled ventilation will be allowed if patient will develop at least one of the following conditions:

* PSV support >20 cmH2O;
* PEEP ≥15 cmH2O;
* unstable hemodynamic status (SBP <90 mmHg with vasoactive drug);
* active cardiac ischemia (dynamic ST changes on cardiac monitor or electrocardiogram);
* unstable arrhythmias (heart rate >140 or <40);
* uncontrolled hypertension (SBP>180 mmHg);
* abrupt decrease in the level of consciousness (RASS <-3);
* dangerous agitation (RASS >+2);
* pH <7.30;
* PaO2/FiO2 ratio ≤100 mmHg;
* necessity to perform diagnostic test (e.g., CT scan or bronchoscopy).

Controlled ventilation will be set on volume mode with Vt 6-8 ml/kg PBW, RR to control pH, unchanged PEEP and FiO2. Controlled ventilation will be thereafter adjusted according to clinical evolution. Patients switched to controlled ventilation will be reassessed at least every 8 hours and they will be switched back to PSV or PSV+Sigh (to maintain study group assignment) targeting the abovementioned settings and adjustments as soon as all the following conditions will be met:

* Patient is able to trigger ventilator breaths;
* PaO2/FiO2 >100 mmHg;
* PEEP <15 cmH2O;
* pH ≥7.3;
* Stable hemodynamic status with stable or decreasing doses of vasopressors for ≥6 hours.

Rescue therapy. In case of desaturation (SpO2 ≤90%) of a patient it will be crucial to exclude hemodynamic impairment as a possible cause. Also, airway obstruction and ventilator malfunction must be ruled out as possible causes. Provided those factors are excluded, a rescue step-up strategy is allowed as follows: institution of protective controlled mechanical ventilation (see above for settings) and performance of recruitment maneuvers at 40-50 cmH2O, PEEP ≥15 cmH2O, prone positioning, inhaled nitric oxide, extracorporeal membrane oxygenation. Patients undergoing rescue treatments will be reassessed at least every 8 hours and switched back to PSV or PSV+Sigh (to maintain study group assignment) with the abovementioned settings and adjustments as soon as all the above mentioned conditions will be met.

Spontaneous breathing trial (SBT). Patients with SpO2 ≥90% on FiO2 ≤0.4 and PEEP ≤5 cmH2O, no agitation, hemodynamically stable with norepinephrine ≤0.1 ug/kg/min or equivalent and at a stable or decreasing dose ≥6 hours and without any of the abovementioned criteria for switch to controlled ventilation will undergo a SBT:

* For patients in the PSV group, the attending physician will perform the SBT directly.
* For patients in the PSV+Sigh group, the attending physician will first withdraw Sigh, wait 60 min and confirm criteria: if confirmed, SBT will be performed; if not, Sigh will be reintroduced and clinical criteria will be checked again to repeat the procedure after at least 8 hours.

SBT will last at least 60 minutes with a combination of PEEP 0-5 cm H2O and PSV 0-5 cm H2O. At the end of the 60 minutes, patient will fail the SBT if any of the following will be present:

* criteria to start the SBT will not be confirmed;
* sustained (>5 min) respiratory rate >35 bpm;
* HR >140 bpm;
* SBP >180 or <80 mmHg;
* marked complaint of dyspnea;
* increased somnolence with elevated pCO2 and/or pH<7.3
* a cough will not be strong enough to clear secretions
* active cardiac ischemia (dynamic ST changes on cardiac monitor or electrocardiogram)
* abrupt decrease in the level of consciousness with RASS <-3. Patients who will fail the SBT will be switched back to PSV or PSV+Sigh (to maintain study group assignment) and clinical criteria will be checked again to repeat the procedure after at least 6 hours.

Patients who will pass the SBT will be extubated or, in the presence of tracheostomy, mechanical ventilation will be discontinued. If a patient will be re-intubated or mechanically ventilated through a tracheostomy again within 48 hours, PSV or PSV+Sigh (to maintain study group assignment) will be restored. If a patient will remain extubated or separated from the ventilator for >48 hours data collection only will continue.

Reasons for re-intubation. After extubation, re-intubation should be promptly performed if at least one of the following criteria is present:

* cardiac arrest;
* respiratory arrest (respiratory pauses with loss of consciousness or gasping for air);
* respiratory failure with SpO2 <90% and/or RR >35 bpm despite NIV;
* decreased level of consciousness impairing ability to protect airway;
* hemoptysis or hematemesis impairing ability to protect airway;
* abundant secretions that cannot be effectively cleared or are associated with lobar collapse, acidosis, hypoxemia, or change in mental status;
* surgical/invasive procedure requiring sedation/anaesthesia +/- neuromuscular blockade such that patient will no longer be able to sustain unassisted breathing;
* hemodynamic instability with SBP <80 mmHg despite vasoactive drugs.

Data collection

At enrolment. Before the Sigh test, the investigators will anonymously collect patients' demographic information (e.g., age, sex, height, weight), past (e.g., hypertension, chronic medications) and recent (e.g., etiology of the acute respiratory failure, days since intubation) medical history, severity of lung injury (e.g., ventilation setting, arterial blood gases, respiratory system compliance, diagnosis of ARDS) and of systemic diseases (e.g., presence of shock, number of organs failure), ventilation settings (e.g., PEEP, FiO2, PSV level).

After the Sigh test. Then, the investigators will collect SatO2/FiO2 change in response to the pre-randomization Sigh test.

First 24 hours from randomization. In both groups for the first 24 hours the investigators will assess every 4 hours the SpO2/FiO2 ratio, RR and tidal volume delivered both during protective PSV and during Sigh to further characterize physiologic response to Sigh over time.

Daily. From day 1 (i.e., within 24 hours from enrollment) to day 28 or death or discharge from the ICU, the following data will be collected every day between 6:00 and 10:00 in the morning: switch from the allocated treatment to the other study arm for ≥24 hours, reason for switch from the allocated treatment, adverse events (i.e., hemodynamic instability with hypotension with SBP <90 mmHg despite vasoactive drugs; arrhythmias with heart rate <40 or >140 bpm; radiographic evidence of barotrauma with pneumothorax, pneumomediastinum, pneumatocoele, or subcutaneous emphysema), arterial SpO2, arterial and central venous blood gas analyses, numbers of quadrants involved on standard chest X-ray, ventilation settings and pattern (i.e., Sigh pressure level, Sigh tidal volume, PSV level, PSV tidal volume, respiratory rate, PEEP, FiO2, minute ventilation, P0.1, mean airway pressure), switch to controlled ventilation for ≥24 hours, reason for switch to controlled ventilation, use of rescue treatments (i.e., use of PEEP ≥15 cmH2O, prone positioning, inhaled nitric oxide, extracorporeal membrane oxygenation), dosage of sedative agents, RASS value, tracheostomy, patient's comfort through visual analog scale, heart rate, arterial blood pressure, central venous pressure, dosage of vaso-active drugs, cumulative fluid balance, SOFA score, SBT failure in the previous 24 hours, reason for SBT failure, time since extubation or separation from mechanical ventilation, time since re-intubation, reason for re-intubation.

Day 28. At day 28, for all enrolled patients, mortality and ventilator-free days will be collected. Ventilator-free days will be calculated as 28 minus the number of days between intubation and successful extubation or separation from mechanical ventilation for tracheostomized patients (i.e., for ≥48 hours).

ELIGIBILITY:
Inclusion Criteria:

* patients intubated since >24 hours and ≤7 days,
* undergoing PSV since >4 and ≤24 hours,
* PaO2/FiO2 ratio ≤300 mmHg (measured at clinical positive end-expiratory pressure [PEEP] and FiO2 values)
* clinical PEEP ≥5 cmH2O,
* Richmond Agitation-Sedation Scale (RASS) value of -2 to 0

Exclusion Criteria:

* patients with PEEP ≥15 cmH2O;
* PaCO2 >60 mmHg;
* Arterial pH <7.30;
* Age <18 year-old;
* PaO2/FiO2 ratio ≤100 mmHg (measured at clinical PEEP and FiO2 values);
* central nervous system or neuromuscular disorders;
* history of severe chronic obstructive pulmonary disease or fibrosis;
* AHRF fully explained by cardiac failure or fluid overload (e.g., left ventricle ejection fraction ≤40% with no other risk factor);
* impossibility to titrate sedation to desired RASS value of -2 to 0;
* evidence of active air leak from the lung (e.g., pneumothorax);
* cardiovascular instability (e.g., systolic blood pressure [SBP] <90 mmHg despite vasopressors);
* clinical suspect of elevated intracranial pressure;
* extracorporeal support;
* moribund status;
* refusal by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Clinical feasibility of PSV+Sigh vs. standard of carde (PSV) | 2 years
  Feasibility will be assessed by measuring the number of patients in each group experiencing at least one of the following failure criteria:
  * switch to controlled ventilation following presence of predefined criteria;
  * use of PEEP ≥15 cmH2O, prone positioning, inhaled nitric oxide, extracorporeal membrane oxygenation;
  * re-intubation within 48 hours from extubation following predefined criteria.
  Based on previous data, the expected rate of failure in patients undergoing PSV will be 22% and we hypothesize a rate of 15% for patients in the PSV+Sigh group. Furthermore, we assume a non-inferiority of the treatment with PSV+Sigh, with a tolerance of 5%. Thus, a sample size of 258 patients (with 129 patients per study arm) will be sufficient to assess feasibility of the PSV+Sigh strategy in this pilot phase with power of 0.8 and alpha 0.05.

SECONDARY OUTCOMES:
Clinical safety of PSV+Sigh comparing adverse events between 2 groups | 2 years
  Compare incidence of the following adverse events in the 2 study groups:
  * hemodynamic instability with hypotension (i.e., SBP <90 mmHg) despite vasoactive drugs;
  * arrhythmias with heart rate <40 or >140 bpm;
  * radiographic evidence of barotrauma (i.e., pneumothorax, pneumomediastinum, pneumatocoele, or subcutaneous emphysema);
  * new chest tube placement.
Quantification of the prevalence of Sigh responders | 2 years
  Quantification of the prevalence of short- (i.e., within 30 minutes) and long-term (i.e., within 24 hours in the PSV+Sigh group) Sigh responders in respect to improved oxygenation.
Mortality | 2 years
  This analysis will be performed comparing the 2 study groups and in responders
Ventilator-free days | 2 years
  This analysis will be performed comparing the 2 study groups and in responders
Number of days on assisted ventilation until day 28 | 28 days
  This analysis will be performed comparing the 2 study groups and in responders
Patients' comfort by visual analog scale | 2 years
  This analysis will be performed comparing the 2 study groups and in responders

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Mauri, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Laurent Brochard, MD, Principal Investigator — St Michael Hospital, Toronto, Canada
Locations (19):
- Tiantan Hospital, Beijing, China
- France (4):
  - CHU Angers, Angers
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hospital de la croix rousse, Lyon
  - GH Sud Ile-de-France, Melun
- UNIVERSITÄTSKLINIKUM Schleswig-Holstein Campus Kiel, Kiel, Germany
- General hospital of Larissa, Larissa, Greece
- Italy (9):
  - Ospedale di Catanzaro Pugliese Ciaccio, Catanzaro
  - Arcispedale Sant'Anna, Ferrara
  - Ospedale San Martino, Genova
  - Ospedale Maggiore Policlinico Cà Granda, Milan
  - Istituto Clinico Humanitas, Milan
  - Ospedale L. Sacco, Milan
  - Ospedale Niguarda, Milan
  - Ospedale San Gerardo, Monza
  - Ospedale Gemelli, Rome
- Spain (2):
  - Vall d'Hebron, Barcelona
  - Foundacion J Diaz, Madrid
- Barking, Havering and Redbridge Hospital, Romford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Matthay MA, Ware LB, Zimmerman GA. The acute respiratory distress syndrome. J Clin Invest. 2012 Aug;122(8):2731-40. doi: 10.1172/JCI60331. Epub 2012 Aug 1. PMID 22850883
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2014 Mar 6;370(10):980. doi: 10.1056/NEJMc1400293. No abstract available. PMID 24597883
- [Background] Mauri T, Foti G, Zanella A, Bombino M, Confalonieri A, Patroniti N, Bellani G, Pesenti A. Long-term extracorporeal membrane oxygenation with minimal ventilatory support: a new paradigm for severe ARDS? Minerva Anestesiol. 2012 Mar;78(3):385-9. PMID 21617600
- [Background] Ranieri VM, Suter PM, Tortorella C, De Tullio R, Dayer JM, Brienza A, Bruno F, Slutsky AS. Effect of mechanical ventilation on inflammatory mediators in patients with acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1999 Jul 7;282(1):54-61. doi: 10.1001/jama.282.1.54. PMID 10404912
- [Background] Hussain SN, Cornachione AS, Guichon C, Al Khunaizi A, Leite Fde S, Petrof BJ, Mofarrahi M, Moroz N, de Varennes B, Goldberg P, Rassier DE. Prolonged controlled mechanical ventilation in humans triggers myofibrillar contractile dysfunction and myofilament protein loss in the diaphragm. Thorax. 2016 May;71(5):436-45. doi: 10.1136/thoraxjnl-2015-207559. Epub 2016 Mar 31. PMID 27033022
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Kallet RH, Matthay MA. Hyperoxic acute lung injury. Respir Care. 2013 Jan;58(1):123-41. doi: 10.4187/respcare.01963. PMID 23271823
- [Background] Bellani G, Guerra L, Musch G, Zanella A, Patroniti N, Mauri T, Messa C, Pesenti A. Lung regional metabolic activity and gas volume changes induced by tidal ventilation in patients with acute lung injury. Am J Respir Crit Care Med. 2011 May 1;183(9):1193-9. doi: 10.1164/rccm.201008-1318OC. Epub 2011 Jan 21. PMID 21257791
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Background] Foti G, Cereda M, Sparacino ME, De Marchi L, Villa F, Pesenti A. Effects of periodic lung recruitment maneuvers on gas exchange and respiratory mechanics in mechanically ventilated acute respiratory distress syndrome (ARDS) patients. Intensive Care Med. 2000 May;26(5):501-7. doi: 10.1007/s001340051196. PMID 10923722
- [Background] Patroniti N, Foti G, Cortinovis B, Maggioni E, Bigatello LM, Cereda M, Pesenti A. Sigh improves gas exchange and lung volume in patients with acute respiratory distress syndrome undergoing pressure support ventilation. Anesthesiology. 2002 Apr;96(4):788-94. doi: 10.1097/00000542-200204000-00004. PMID 11964584
- [Background] Nacoti M, Spagnolli E, Bonanomi E, Barbanti C, Cereda M, Fumagalli R. Sigh improves gas exchange and respiratory mechanics in children undergoing pressure support after major surgery. Minerva Anestesiol. 2012 Aug;78(8):920-9. Epub 2012 Apr 27. PMID 22531559
- [Background] Mauri T, Eronia N, Abbruzzese C, Marcolin R, Coppadoro A, Spadaro S, Patroniti N, Bellani G, Pesenti A. Effects of Sigh on Regional Lung Strain and Ventilation Heterogeneity in Acute Respiratory Failure Patients Undergoing Assisted Mechanical Ventilation. Crit Care Med. 2015 Sep;43(9):1823-31. doi: 10.1097/CCM.0000000000001083. PMID 25985386
- [Background] Tabuchi A, Nickles HT, Kim M, Semple JW, Koch E, Brochard L, Slutsky AS, Pries AR, Kuebler WM. Acute Lung Injury Causes Asynchronous Alveolar Ventilation That Can Be Corrected by Individual Sighs. Am J Respir Crit Care Med. 2016 Feb 15;193(4):396-406. doi: 10.1164/rccm.201505-0901OC. PMID 26513710
- [Background] Guldner A, Braune A, Carvalho N, Beda A, Zeidler S, Wiedemann B, Wunderlich G, Andreeff M, Uhlig C, Spieth PM, Koch T, Pelosi P, Kotzerke J, de Abreu MG. Higher levels of spontaneous breathing induce lung recruitment and reduce global stress/strain in experimental lung injury. Anesthesiology. 2014 Mar;120(3):673-82. doi: 10.1097/ALN.0000000000000124. PMID 24406799
- [Background] Moraes L, Santos CL, Santos RS, Cruz FF, Saddy F, Morales MM, Capelozzi VL, Silva PL, de Abreu MG, Garcia CS, Pelosi P, Rocco PR. Effects of sigh during pressure control and pressure support ventilation in pulmonary and extrapulmonary mild acute lung injury. Crit Care. 2014 Aug 12;18(4):474. doi: 10.1186/s13054-014-0474-4. PMID 25113136
- [Background] Goligher EC, Kavanagh BP, Rubenfeld GD, Ferguson ND. Physiologic Responsiveness Should Guide Entry into Randomized Controlled Trials. Am J Respir Crit Care Med. 2015 Dec 15;192(12):1416-9. doi: 10.1164/rccm.201410-1832CP. PMID 25580530
- [Background] Riker RR, Fugate JE; Participants in the International Multi-disciplinary Consensus Conference on Multimodality Monitoring. Clinical monitoring scales in acute brain injury: assessment of coma, pain, agitation, and delirium. Neurocrit Care. 2014 Dec;21 Suppl 2:S27-37. doi: 10.1007/s12028-014-0025-5. PMID 25208671
- [Background] Goligher EC, Kavanagh BP, Rubenfeld GD, Adhikari NK, Pinto R, Fan E, Brochard LJ, Granton JT, Mercat A, Marie Richard JC, Chretien JM, Jones GL, Cook DJ, Stewart TE, Slutsky AS, Meade MO, Ferguson ND. Oxygenation response to positive end-expiratory pressure predicts mortality in acute respiratory distress syndrome. A secondary analysis of the LOVS and ExPress trials. Am J Respir Crit Care Med. 2014 Jul 1;190(1):70-6. doi: 10.1164/rccm.201404-0688OC. PMID 24919111
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Xirouchaki N, Kondili E, Vaporidi K, Xirouchakis G, Klimathianaki M, Gavriilidis G, Alexandopoulou E, Plataki M, Alexopoulou C, Georgopoulos D. Proportional assist ventilation with load-adjustable gain factors in critically ill patients: comparison with pressure support. Intensive Care Med. 2008 Nov;34(11):2026-34. doi: 10.1007/s00134-008-1209-2. Epub 2008 Jul 8. PMID 18607562
- [Result] Peek GJ, Mugford M, Tiruvoipati R, Wilson A, Allen E, Thalanany MM, Hibbert CL, Truesdale A, Clemens F, Cooper N, Firmin RK, Elbourne D; CESAR trial collaboration. Efficacy and economic assessment of conventional ventilatory support versus extracorporeal membrane oxygenation for severe adult respiratory failure (CESAR): a multicentre randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1351-63. doi: 10.1016/S0140-6736(09)61069-2. Epub 2009 Sep 15. PMID 19762075
- [Derived] Rezoagli E, Fornari C, Fumagalli R, Grasselli G, Volta CA, Navalesi P, Knafelj R, Brochard L, Pesenti A, Mauri T, Foti G; Pleural Pressure Working Group (PLUG). Heterogeneous impact of Sighs on mortality in patients with acute hypoxemic respiratory failure: insights from the PROTECTION study. Ann Intensive Care. 2024 Oct 5;14(1):153. doi: 10.1186/s13613-024-01385-0. PMID 39368033
- [Derived] Mauri T, Foti G, Fornari C, Grasselli G, Pinciroli R, Lovisari F, Tubiolo D, Volta CA, Spadaro S, Rona R, Rondelli E, Navalesi P, Garofalo E, Knafelj R, Gorjup V, Colombo R, Cortegiani A, Zhou JX, D'Andrea R, Calamai I, Vidal Gonzalez A, Roca O, Grieco DL, Jovaisa T, Bampalis D, Becher T, Battaglini D, Ge H, Luz M, Constantin JM, Ranieri M, Guerin C, Mancebo J, Pelosi P, Fumagalli R, Brochard L, Pesenti A; PROTECTION Trial Collaborators. Sigh in Patients With Acute Hypoxemic Respiratory Failure and ARDS: The PROTECTION Pilot Randomized Clinical Trial. Chest. 2021 Apr;159(4):1426-1436. doi: 10.1016/j.chest.2020.10.079. Epub 2020 Nov 13. PMID 33197403
- [Derived] Mauri T, Foti G, Fornari C, Constantin JM, Guerin C, Pelosi P, Ranieri M, Conti S, Tubiolo D, Rondelli E, Lovisari F, Fossali T, Spadaro S, Grieco DL, Navalesi P, Calamai I, Becher T, Roca O, Wang YM, Knafelj R, Cortegiani A, Mancebo J, Brochard L, Pesenti A; Protection Study Group. Pressure support ventilation + sigh in acute hypoxemic respiratory failure patients: study protocol for a pilot randomized controlled trial, the PROTECTION trial. Trials. 2018 Aug 29;19(1):460. doi: 10.1186/s13063-018-2828-8. PMID 30157955